CLINICAL TRIAL: NCT06191159
Title: A Randomized Controlled Trial Comparing the Cosmetic Outcome of Electrocautery, Scalpel and PEAK PlasmaBlade for Surgical Breast Incisions
Brief Title: Cosmetic Outcome of Electrocautery, Scalpel and PEAK PlasmaBlade for Surgical Breast Incisions
Acronym: SCPPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Carol Dingee, Breast Surgical Oncologist, Principal Investigator, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H23-00115
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Wound Complication; Surgical Wound Infection; Post-operative Pain; Postoperative Complications; Scar
Keywords: Electrocautery; PEAK PlasmaBlade; Scalpel; Mastectomy; Incision
MeSH Terms: conditions — Surgical Wound Infection; Pain, Postoperative; Postoperative Complications; Cicatrix; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in equal numbers to have the initial skin incision made with either scalpel, standard electrocautery or PEAK PlasmaBlade. For skin incisions made with electrocautery or PEAK PlasmaBlade the surgeon will use the same equipment for the completion of the surgery. Patients who have initial skin incision with scalpel will be further randomized to have completion of the surgery with standard electrocautery or PEAK PlasmaBlade. Any patients with bilateral mastectomy will be randomized to the same surgical approach for both breasts.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (Active Comparator): The Standard of Care arm will consist of the scalpel for the initial skin incision and further randomization to have completion of the surgery with standard electrocautery or PEAK PlasmaBlade.
  Interventions: Device: Scalpel and standard electrocautery or PEAK PlasmaBlade
- PEAK PlasmaBlade (Experimental): The PEAK PlasmaBlade will be used for the entirety of the surgery, including the initial skin incision.
  Interventions: Device: PEAK PlasmaBlade
- Standard Electrocautery (Experimental): Standard electrocautery will be used for the entirety of the surgery, including the initial skin incision.
  Interventions: Device: Standard Electrocautery

INTERVENTIONS:
Device: Scalpel and standard electrocautery or PEAK PlasmaBlade — Scalpel followed by completion of surgery with standard electrocautery or PEAK PlasmaBlade.
  Arms: Standard of Care
Device: PEAK PlasmaBlade — PEAK PlasmaBlade for entire surgery.
  Arms: PEAK PlasmaBlade
Device: Standard Electrocautery — Standard Electrocautery for entire surgery.
  Arms: Standard Electrocautery

SUMMARY:
This study will compare the cosmetic scar result from the use of scalpel, electrocautery, and pulsed electron avalanche knife (PEAK) PlasmaBlade (PPB) for the initial skin incision for total mastectomy procedures without immediate breast reconstruction.

It is hypothesized that there will be no significant difference in mastectomy scar cosmesis.

The purpose and objectives of this study are:

1. To evaluate and compare the cosmetic scar result from the use of scalpel, standard electrocautery, or PEAK PlasmaBlade for initial incision for total mastectomy procedures without immediate breast reconstruction.
2. To inform future equipment choices for breast surgery including potential elimination of scalpels and their attendant risks.

DETAILED DESCRIPTION:
Scalpel, electrocautery, and PEAK PlasmaBlade (PPB) have all been shown to be safe techniques for surgical incision, but no study has proven the superiority for cosmesis for PPB incision when compared to conventional electrocautery or scalpel.

The investigators propose a double blind prospective randomized controlled study of consecutive patients scheduled for total mastectomy +/- axilla staging without immediate breast reconstruction to evaluate the cosmetic scar result from the use of scalpel, standard electrocautery or PEAK PlasmaBlade.

Scar cosmesis will be evaluated postoperatively at two-to-four weeks, six months, and twelve months by two independent observers blinded to the equipment used, and patient reported outcomes will be reported using the validated SCAR-Q questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a total mastectomy with or without axilla surgical staging

Exclusion Criteria:

* Patients having immediate breast reconstruction
* Patients with a diagnosis of inflammatory breast cancer
* History of keloid scar formation
* History of connective tissue disorder (scleroderma or rheumatoid arthritis with skin involvement)
* Patients with prior incision at the planned mastectomy site.
* Patients with known suture hypersensitivity
* Patients with evidence of current infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Scar cosmesis (SCAR scale) | 2-4 weeks post-operatively
  Mastectomy site scar cosmesis will be evaluated 2-4 weeks post-operatively by two independent observers blinded to the equipment used for the surgery using photo evaluation with the Scar Cosmesis Assessment and Rating (SCAR) scale. The SCAR scale yields scores ranging from a minimum score of 0 (best possible scar) to a maximum score of 15 (worst possible scar).
Scar cosmesis (Vancouver Scar Scale) | 2-4 weeks post-operatively
  Mastectomy site scar cosmesis will be evaluated 2-4 weeks post-operatively by the treating surgeon using the Vancouver Scar Scale for physical examination. The Vancouver Scar Scale yields scores ranging from 0 (best) to 13 (worst).
Scar cosmesis (SCAR-Q) | 2-4 weeks post-operatively
  Patient reported outcomes will be reported 2-4 weeks post-operatively using the SCAR-Q scale, a comprehensive scar appearance scale with independently functioning domains for scar appearance, scar symptoms and psychosocial impact, which each yield transformed scores ranging from 0 (worst) to 100 (best).
Scar cosmesis (SCAR scale) | 6 months post-operatively
  Mastectomy site scar cosmesis will be evaluated 6 months post-operatively by two independent observers blinded to the equipment used for the surgery using photo evaluation with the Scar Cosmesis Assessment and Rating (SCAR) scale. The SCAR scale yields scores ranging from a minimum score of 0 (best possible scar) to a maximum score of 15 (worst possible scar).
Scar cosmesis (Vancouver Scar Scale) | 6 months post-operatively
  Mastectomy site scar cosmesis will be evaluated 6 months post-operatively by the treating surgeon using the Vancouver Scar Scale for physical examination. The Vancouver Scar Scale yields scores ranging from 0 (best) to 13 (worst).
Scar cosmesis (SCAR-Q) | 6 months post-operatively
  Patient reported outcomes will be reported 6 months post-operatively using the SCAR-Q scale, a comprehensive scar appearance scale with independently functioning domains for scar appearance, scar symptoms and psychosocial impact, which each yield transformed scores ranging from 0 (worst) to 100 (best).
Scar cosmesis (SCAR scale) | 12 months post-operatively
  Mastectomy site scar cosmesis will be evaluated 12 months post-operatively by two independent observers blinded to the equipment used for the surgery using photo evaluation with the Scar Cosmesis Assessment and Rating (SCAR) scale. The SCAR scale yields scores ranging from a minimum score of 0 (best possible scar) to a maximum score of 15 (worst possible scar).
Scar cosmesis (Vancouver Scar Scale) | 12 months post-operatively
  Mastectomy site scar cosmesis will be evaluated 12 months post-operatively by the treating surgeon using the Vancouver Scar Scale for physical examination. The Vancouver Scar Scale yields scores ranging from 0 (best) to 13 (worst).
Scar cosmesis (SCAR-Q) | 12 months post-operatively
  Patient reported outcomes will be reported 12 months post-operatively using the SCAR-Q scale, a comprehensive scar appearance scale with independently functioning domains for scar appearance, scar symptoms and psychosocial impact, which each yield transformed scores ranging from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Development of post-operative seroma | within 12 months post-operatively
  Development of post-operative seroma, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Development of post-operative hematoma | within 12 months post-operatively
  Development of post-operative hematoma, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Development of excessive bruising | within 12 months post-operatively
  Development of post-operative excessive bruising, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Development of flap necrosis | within 12 months post-operatively
  Development of post-operative flap-necrosis, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Development of wound dehiscence | within 12 months post-operatively
  Development of post-operative wound dehiscence, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Development of cellulitis | within 12 months post-operatively
  Development of post-operative cellulitis, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Delayed healing | within 12 months post-operatively
  Delayed healing post-operatively, graded using the Clavien-Dindo classification system for surgical complications. The Clavien-Dindo classification of surgical complications ranges from Grade I (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions) to Grade V (death of a patient).
Wound infection rate | within 12 months post-operatively
  Development of wound infection post-operatively.
Length of operative procedure | beginning to end of operative procedure
  The duration of the operative procedure.
Intraoperative blood loss | beginning to end of operative procedure
  Volume of blood loss during the operative procedure.
Peri-operative pain | from end of operative procedure to 2 weeks post-operatively
  Peri-operative pain will be indicated by the medication prescribed and/or taken during post-anesthesia recovery (PAR) and surgical daycare.
Duration of drain | from drain placement to drain removal, up to 1 month
  The total time between drain placement and removal. Drain removal will occur when less than 30 mL of drainage accumulates for two consecutive days.
Volume of measured drainage | from drain placement to drain removal, up to 1 month
  Volume of drainage measured throughout drain duration. Drain removal will occur when less than 30 mL of drainage accumulates for two consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Carol K Dingee, MD, FRCSC, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- Mount Saint Joseph Hospital, Vancouver, British Columbia, Canada